CLINICAL TRIAL: NCT06946004
Title: The Potential of Normobaric Oxygen Therapy to Enhance Erythropoiesis, Reduce Oxidative Stress, and Modulate Immune Function in Colorectal Cancer Patients Undergoing Chemotherapy: Study Protocol for a Prospective, Randomized, Double-Blind, Placebo-Controlled Trial (NBO-ONCO)
Brief Title: Normobaric Oxygen Therapy in Colorectal Cancer Patients
Acronym: NBO-ONCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Collaborators: Wroclaw Medical University (Poland) (Unknown); Wroclaw University of Science and Technology (Poland) (Unknown); Hirszfeld Institute of Immunology and Experimental Therapy, Polish Academy of Sciences (Poland) (Unknown); WSB Merito University in Opole (Poland) (Unknown); Academy of Applied Sciences in Nowy Sacz (Poland) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024/ABM/02/00007
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer (CRC)
Keywords: colorectal cancer; normobaric oxygen therapy; chemotherapy-induced anemia; oxidative stress; immune modulation; erythropoiesis; supportive cancer care; adverse effects; stress; anxiety; depression; psychological well-being; quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded, ensuring that neither patients nor the research team involved in data analysis know the allocation to active or placebo NBO, preserving objectivity in outcome assessment. Patients and clinical staff (excluding NBO operators who administer the therapy) are blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active NBO therapy (n=127) (Experimental): Patient's exposure to NBO conditions in group 1 (aNBO)
  Interventions: Device: Normobaric oxygen therapy
- placebo NBO therapy (n=127) (Placebo Comparator): Patients' exposure to atmospheric conditions in the same NBO chamber without normobaric conditions in group 2 (pNBO)
  Interventions: Device: Normobaric oxygen therapy

INTERVENTIONS:
Device: Normobaric oxygen therapy — Patient's exposure to NBO conditions in group 1 (aNBO) including: oxygen levels of 32-40% (compared to about 21% in the atmosphere), pressure maintained at 1,500 hPa (about 1,000 hPa outside), carbon dioxide levels between 0.7-1.9% (compared to 0.03% in the atmosphere, and hydrogen levels between 0.5-1% (which is 10 to 20 thousand times higher than in the atmosphere). Exposure time in the NBO chamber will be the standard 2 hours with an additional 20 minutes for preparation and adaptation and 10 minutes for finalization and the decompression period.
  Arms: active NBO therapy (n=127)
Device: Normobaric oxygen therapy — Patients' exposure to atmospheric conditions in the same NBO chamber (without normobaric conditions to provide placebo intervention as the study comparator) in group 2 (pNBO): oxygen levels about 21%, pressure maintained at about 1,000 hPa, carbon dioxide levels about o 0.03%, and hydrogen levels about 0.00005% (0.5 parts per million, like in the atmos-phere).
  Arms: placebo NBO therapy (n=127)

SUMMARY:
Colorectal cancer (CRC) patients undergoing chemotherapy often experience anemia, oxidative stress, and immune suppression, significantly impacting their quality of life and treatment outcomes. Normobaric oxygen (NBO) therapy, which delivers oxygen at atmospheric pressure with elevated oxygen concentration, has shown a potential to enhance erythropoiesis, reduce oxidative stress, and modulate immune function. However, its efficacy in CRC patients remains underexplored. This study aims to evaluate the effects of NBO exposures on (1) supporting erythropoiesis by measuring erythropoietin (EPO) levels and hypoxia-inducible factors (HIF-1α), (2) reducing oxidative stress and improving stress and emotional well-being, and (3) modulating immune function by assessing cytokine profiles. Secondary objectives include assessing the impact of NBO on patient-reported outcome measures (PROMs) such as stress, anxiety, depression, and quality of life. This is a prospective, randomized, double-blind, placebo-controlled clinical trial. A total of 254 CRC patients undergoing chemotherapy will be randomized 1:1 to receive either active NBO therapy (n=127) or placebo NBO therapy (n=127). The intervention consists of 10 NBO sessions over five weeks. Primary outcomes include biomarkers of erythropoiesis, oxidative stress, and immune response. Secondary outcomes assess quality of life and psychological well-being. Data will be collected at baseline, mid-intervention, post-intervention, and during two follow-up visits (3- and 6-months post-intervention). The study hypothesizes that NBO therapy will improve erythropoiesis, reduce oxidative stress, and enhance immune function in CRC patients, leading to improved quality of life and clinical outcomes. Findings from this trial may establish NBO as a novel supportive therapy for CRC patients undergoing chemotherapy.

DETAILED DESCRIPTION:
The intervention will involve NBO as a supportive treatment for CRC patients undergoing chemotherapy. The NBO protocol consists of regular sessions in a normobaric chamber where patients are exposed to controlled oxygen levels aimed at reducing ox-idative stress, supporting erythropoiesis, and modulating immune function. Patients in the CRC group will undergo 10 NBO sessions across five weeks, with two sessions weekly.

Patient's exposure to NBO conditions in group 1 (aNBO) including: oxygen levels of 32-40% (compared to about 21% in the atmosphere), pressure maintained at 1,500 hPa (about 1,000 hPa outside), carbon dioxide levels between 0.7-1.9% (compared to 0.03% in the atmosphere, and hydrogen levels between 0.5-1% (which is 10 to 20 thousand times higher than in the atmosphere). Exposure time in the NBO chamber will be the standard 2 hours with an additional 20 minutes for preparation and adaptation and 10 minutes for the finalization and decompression period.

Patients' exposure to atmospheric conditions in the same NBO chamber (without normobaric conditions to provide sham-placebo intervention) in group 2 (pNBO): oxygen levels about 21%, pressure maintained at about 1,000 hPa, carbon dioxide levels about o 0.03%, and hydrogen levels about 0.00005% (0.5 parts per million, like in the atmos-phere). The primary comparator in this study is the placebo NBO group (CRC patients; n=127) for CRC patients, which serves to differentiate the specific effects of active NBO from the natural course of treatment without enhanced oxygen exposure.

The patient assessment scheme contains six visits from V0 to V5 with subsequent analytical packages with detailed explanation in 2.8. section. The patient assessment schedule consists of six visits, from V0 to V5, each including specific evaluations and interventions. The study begins with V0 (prequalification/screening), where patient consent is obtained, medical history is collected, and baseline data are recorded. V1 (randomization and pre-test visit) involves the initial assessments, including anemia, stress, immune, genetic markers, and patient-reported outcomes (PROMs). Following this, the first phase of the NBO intervention (sessions 1-5) takes place over five weeks. At V2 (midpoint evaluation), the same set of assessments is repeated to track progress, followed by the second phase of the NBO intervention (sessions 6-10) conducted over the next five weeks. V3 (finalization and post-test visit) marks the completion of the intervention, with a final round of primary and secondary outcome assessments. The study then proceeds with two follow-up visits: V4 (3-months post-NBO) and V5 (6-months post-NBO), where anemia, stress, immune, genetic markers, and PROMs are reassessed to evaluate the long-term effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years (participants must be adults)
* diagnosed with CRC (stage II-IV, scheduled for standard chemotherapy (for study and control groups)
* baseline hemoglobin levels above 10 g/dL
* no concurrent hematologic malignancies
* eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (ensuring participants are ambulatory and capable of self-care)
* life expectancy of at least 12 months (participants are expected to survive the duration of the study)
* ability and willingness to comply with all study procedures and schedules (including NBO therapy sessions and follow-up visits)
* adequate organ function as determined by laboratory tests (liver function tests - ALT, AST), renal function tests (serum creatinine, eGFR)
* women of childbearing potential must have a negative pregnancy test prior to enrollment and agree to use effective contraception during the study (to ensure safety for potential pregnancies)
* written informed consent obtained prior to any study-related procedures (participants must understand and agree to all aspects of the study).

Exclusion Criteria:

* age under 18 years or over 80 years
* severe cardiovascular or respiratory conditions (e.g., unstable angina, recent myocardial infarction, advanced COPD)
* severe anemia (hemoglobin <10 g/dL) or any hemolytic disorder that could confound study outcomes
* uncontrolled diabetes mellitus (e.g., HbA1c >8.0% or poor glycemic control requiring frequent hospitalizations)
* pregnancy or breastfeeding
* severe infection or immunocompromised status unrelated to cancer (e.g., advanced HIV infection)
* current psychiatric or neurological disorders that could interfere with study participation
* participation in other investigational therapies within the last 30 days; (9) lack of written informed consent for study participation
* autoimmune or inflammatory conditions (e.g., lupus, rheumatoid arthritis on immunosuppressive therapy) that significantly alter immune responses
* presence of any contraindication for NBO therapy (e.g., active bleeding, acute infections, inflammation of the optic nerve, epilepsy or seizures, uncontrolled diabetes as noted above, pneumothorax, emphysema, electronic implants).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Erythropoietin (EPO) concentration | From enrollment to the end of 6th month follow-up
  Erythropoietin (EPO) concentration [mU/mL] will be measured using a quantitative immunoassay (ELISA) at V1, V2, V3, V4, and V5.
Hypoxia-inducible factor-1α (HIF-1α) | From enrollment to the end of 6th month follow-up
  Hypoxia-inducible factor-1α (HIF-1α) [ng/mL] will be measured using a quantitative immunoassay at V1, V2, V3, V4, and V5.
Reticulocyte count | From enrollment to the end of 6th month follow-up
  Reticulocyte count [% of total red blood cells] will be measured using an automated hematology analyzer at V1, V2, V3, V4, and V5.
Red blood cell (RBC) | From enrollment to the end of 6th month follow-up
  Red blood cell (RBC) count [10¹² cells/L] will be measured using 5-part differential blood morphology on an automated hematology analyzer at V1, V2, V3, V4, and V5.
Hemoglobin concentration (HGB) | From enrollment to the end of 6th month follow-up
  Hemoglobin concentration (HGB) [g/dL] will be measured using an automated hematology analyzer at V1, V2, V3, V4, and V5.
Hematocrit | From enrollment to the end of 6th month follow-up
  Hematocrit [%] will be measured using an automated hematology analyzer at V1, V2, V3, V4, and V5.
Serum creatinine | From enrollment to the end of 6th month follow-up
  Serum creatinine [µmol/L] will be measured using an enzymatic assay at V1, V2, V3, V4, and V5.
Estimated glomerular filtration rate (eGFR) | From enrollment to the end of 6th month follow-up
  Estimated glomerular filtration rate (eGFR) [mL/min/1.73 m²] will be calculated using the CKD-EPI equation at V1, V2, V3, V4, and V5.
Alanine aminotransferase (ALT) | From enrollment to the end of 6th month follow-up
  Alanine aminotransferase (ALT) [IU/L] will be measured using an enzymatic assay at V1, V2, V3, V4, and V5.
Aspartate aminotransferase (AST) | From enrollment to the end of 6th month follow-up
  Aspartate aminotransferase (AST) [IU/L] will be measured using an enzymatic assay at V1, V2, V3, V4, and V5.
Fasting glucose | From enrollment to the end of 6th month follow-up
  Fasting glucose [mmol/L] will be measured using a hexokinase assay at V1, V2, V3, V4, and V5.
Fasting insulin | From enrollment to the end of 6th month follow-up
  Fasting insulin [µU/mL] will be measured using an immunoassay at V1, V2, V3, V4, and V5.
Lipid profile | From enrollment to the end of 6th month follow-up
  Lipid profile (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides) [mmol/L] will be measured using enzymatic/colorimetric assays at V1, V2, V3, V4, and V5.
Iron metabolism (serum iron, total iron-binding capacity [TIBC] | From enrollment to the end of 6th month follow-up
  Iron metabolism (serum iron, total iron-binding capacity [TIBC] [µmol/L], ferritin [ng/mL], vitamin B₁₂ [pg/mL]) will be measured using immunoassays at V1, V2, V3, V4, and V5.
Serum albumin | From enrollment to the end of 6th month follow-up
  Serum albumin [g/L] will be measured using a bromcresol green assay at V1, V2, V3, V4, and V5.
C-reactive protein (CRP) | From enrollment to the end of 6th month follow-up
  C-reactive protein (CRP) [mg/L] will be measured using a high-sensitivity immunoturbidimetric assay at V1, V2, V3, V4, and V5.
Reactive oxygen species (ROS) level | From enrollment to the end of 6th month follow-up]
  Reactive oxygen species (ROS) level [relative fluorescence units] will be measured using a chemiluminescence assay at V1, V2, V3, V4, and V5.
Serum cortisol | From enrollment to the end of 6th month follow-up
  Serum cortisol [µg/dL] will be measured using a high-sensitivity immunoassay at V1, V2, V3, V4, and V5.
Gamma-aminobutyric acid (GABA) | From enrollment to the end of 6th month follow-up
  Gamma-aminobutyric acid (GABA) [µmol/L] will be measured using an enzyme-linked immunosorbent assay at V1, V2, V3, V4, and V5.
Dopamine | From enrollment to the end of 6th month follow-up
  Dopamine [ng/mL] will be measured using a competitive immunoassay at V1, V2, V3, V4, and V5.
Serotonin | From enrollment to the end of 6th month follow-up
  Serotonin [ng/mL] will be measured using a competitive immunoassay at V1, V2, V3, V4, and V5.
Fibrinogen | From enrollment to the end of 6th month follow-up
  Fibrinogen [g/L] will be measured using the Clauss clotting assay at V1, V2, V3, V4, and V5.
Glycated hemoglobin (HbA₁c) | From enrollment to the end of 6th month follow-up
  Glycated hemoglobin (HbA₁c) [%] will be measured using high-performance liquid chromatography at V1, V2, V3, V4, and V5.
Dehydroepiandrosterone-sulfate (DHEA-S) | From enrollment to the end of 6th month follow-up
  Dehydroepiandrosterone-sulfate (DHEA-S) [µg/dL] will be measured using an immunoassay at V1, V2, V3, V4, and V5.
Systolic blood pressure (SBP) | From enrollment to the end of 6th month follow-up
  Systolic blood pressure (SBP) [mmHg] will be measured using an automated sphygmomanometer at V1, V2, V3, V4, and V5.
Diastolic blood pressure (DBP) | From enrollment to the end of 6th month follow-up
  Diastolic blood pressure (DBP) [mmHg] will be measured using an automated sphygmomanometer at V1, V2, V3, V4, and V5.
Heart rate (HR) | From enrollment to the end of 6th month follow-up
  Heart rate (HR) [beats per minute] will be measured using an automated sphygmomanometer at V1, V2, V3, V4, and V5.
Body mass index (BMI) | From enrollment to the end of 6th month follow-up
  Body mass index (BMI) [kg/m²] will be calculated from measured weight and height at V1, V2, V3, V4, and V5.
Body surface area (BSA) | From enrollment to the end of 6th month follow-up
  Body surface area (BSA) [m²] will be calculated using the Mosteller formula from measured weight and height at V1, V2, V3, V4, and V5.
Waist-to-hip ratio (WHR) | From enrollment to the end of 6th month follow-up
  Waist-to-hip ratio (WHR) [ratio] will be calculated from measured waist and hip circumferences at V1, V2, V3, V4, and V5.
Tumor necrosis factor-α (TNF-α) | From enrollment to the end of 6th month follow-up
  Tumor necrosis factor-α (TNF-α) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Interleukin-1β (IL-1β) | From enrollment to the end of 6th month follow-up
  Interleukin-1β (IL-1β) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Interleukin-6 (IL-6) | From enrollment to the end of 6th month follow-up
  Interleukin-6 (IL-6) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Interleukin-10 (IL-10) | From enrollment to the end of 6th month follow-up
  Interleukin-10 (IL-10) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Monocyte chemoattractant protein-1 (MCP-1/CCL2) | From enrollment to the end of 6th month follow-up
  Monocyte chemoattractant protein-1 (MCP-1/CCL2) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Macrophage inflammatory protein-1α (MIP-1α/CCL3) | From enrollment to the end of 6th month follow-up
  Macrophage inflammatory protein-1α (MIP-1α/CCL3) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Macrophage inflammatory protein-1β (MIP-1β/CCL4) | From enrollment to the end of 6th month follow-up
  Macrophage inflammatory protein-1β (MIP-1β/CCL4) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Vascular endothelial growth factor A (VEGF-A) | From enrollment to the end of 6th month follow-up
  Vascular endothelial growth factor A (VEGF-A) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.
Platelet-derived growth factor-BB (PDGF-BB) | From enrollment to the end of 6th month follow-up
  Platelet-derived growth factor-BB (PDGF-BB) [pg/mL] will be measured using a multiplex immunoassay (Luminex) at V1, V2, V3, V4, and V5.

SECONDARY OUTCOMES:
Stress level (self-assessment) | From enrollment to the end of 6th month follow-up
  The Perceived Stress Questionnaire (PSQ-30) is a 30-item self-report instrument designed to assess perceived stress over the previous month. Each item is rated on a 4-point Likert scale (1 = "almost never" to 4 = "usually"), yielding a raw score that can range from 30 (minimum) to 120 (maximum). Higher raw scores indicate greater perceived stress (worse outcome). The PSQ-30 will be administered at V1, V2, V3, V4, and V5.
Anxiety and depression levels (self-assessment) | From enrollment to the end of 6th month follow-up
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire comprising two subscales: HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D). Each subscale contains 7 items scored on a 4-point Likert scale (0 = "not at all" to 3 = "very often"), yielding subscale scores from 0 (minimum) to 21 (maximum). Higher scores indicate greater symptom severity (worse outcome). The HADS total score (sum of HADS-A and HADS-D) ranges from 0 to 42. The HADS will be administered at V1, V2, V3, V4, and V5.
Quality of live level (self-assessment) | From enrollment to the end of 6th month follow-up
  EuroQol Five-Dimension Five-Level questionnaire (EQ-5D-5L) index score [-0.59 to 1.00; higher = better health] will be derived from five domains-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated on a 5-point scale (1 = no problems to 5 = extreme problems). Health states will be converted to a single index value using the Polish EQ-5D-5L value set. The EQ-5D-5L will be administered at V1, V2, V3, V4, and V5.

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Military Clinical Hospital, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin CH, Su WH, Chen YC, Feng PH, Shen WC, Ong JR, Wu MY, Wong CS. Treatment with normobaric or hyperbaric oxygen and its effect on neuropsychometric dysfunction after carbon monoxide poisoning: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Sep;97(39):e12456. doi: 10.1097/MD.0000000000012456. PMID 30278526
- [Background] Bloch Y, Belmaker RH, Shvartzman P, Romem P, Bolotin A, Bersudsky Y, Azab AN. Normobaric oxygen treatment for mild-to-moderate depression: a randomized, double-blind, proof-of-concept trial. Sci Rep. 2021 Sep 23;11(1):18911. doi: 10.1038/s41598-021-98245-9. PMID 34556722
- [Background] Kujawski S, Slomko J, Morten KJ, Murovska M, Buszko K, Newton JL, Zalewski P. Autonomic and Cognitive Function Response to Normobaric Hyperoxia Exposure in Healthy Subjects. Preliminary Study. Medicina (Kaunas). 2020 Apr 10;56(4):172. doi: 10.3390/medicina56040172. PMID 32290164
- [Background] De Bels D, Theunissen S, Devriendt J, Germonpre P, Lafere P, Valsamis J, Snoeck T, Meeus P, Balestra C. The 'normobaric oxygen paradox': does it increase haemoglobin? Diving Hyperb Med. 2012 Jun;42(2):67-71. PMID 22828812
- [Background] Saleh EAM, Al-Dolaimy F, Qasim Almajidi Y, Baymakov S, Kader M MA, Ullah MI, Abbas AHR, Khlewee IH, Bisht YS, Alsaalamy AH. Oxidative stress affects the beginning of the growth of cancer cells through a variety of routes. Pathol Res Pract. 2023 Sep;249:154664. doi: 10.1016/j.prp.2023.154664. Epub 2023 Jul 1. PMID 37573621
- [Background] Noman MZ, Hasmim M, Lequeux A, Xiao M, Duhem C, Chouaib S, Berchem G, Janji B. Improving Cancer Immunotherapy by Targeting the Hypoxic Tumor Microenvironment: New Opportunities and Challenges. Cells. 2019 Sep 14;8(9):1083. doi: 10.3390/cells8091083. PMID 31540045
- [Background] Bozzini C, Busti F, Marchi G, Vianello A, Cerchione C, Martinelli G, Girelli D. Anemia in patients receiving anticancer treatments: focus on novel therapeutic approaches. Front Oncol. 2024 Apr 2;14:1380358. doi: 10.3389/fonc.2024.1380358. eCollection 2024. PMID 38628673
- [Background] Bray F, Jemal A, Grey N, Ferlay J, Forman D. Global cancer transitions according to the Human Development Index (2008-2030): a population-based study. Lancet Oncol. 2012 Aug;13(8):790-801. doi: 10.1016/S1470-2045(12)70211-5. Epub 2012 Jun 1. PMID 22658655
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338